CLINICAL TRIAL: NCT03014726
Title: ROBUST I Pilot Study, ROBUST I Study, Re-Establishing Flow Via Drug Coated Balloon For The Treatment Of Urethral Stricture Disease
Brief Title: ROBUST I Pilot Study, Re-Establishing Flow Via Drug Coated Balloon For The Treatment Of Urethral Stricture Disease
Acronym: ROBUST
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC016
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Stricture Urethra
Keywords: reduced urine flow rate; low peak flow rate; urinary tract infections
MeSH Terms: conditions — Urethral Stricture; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DCB Treatment (Experimental): Stricture patients treated by DCB
  Interventions: Combination Product: Urotronic Drug Coated Balloon (DCB)

INTERVENTIONS:
Combination Product: Urotronic Drug Coated Balloon (DCB) — Urotronic Drug Coated Balloon (DCB) is a catheter with a tapered atraumatic tip. The distal end of the catheter has a semi-compliant inflatable balloon coated with a proprietary coating containing the drug and carriers.

SUMMARY:
Robust I study is a feasibility study for evaluating the safety and efficacy of DCB.

DETAILED DESCRIPTION:
The study is designed to determine the safety and effectiveness for drug coated balloon (DCB).

Up to 50 subjects is planned to be enrolled and treated with the study device at up to 5 clinical sites outside of US. Due to significantly higher prevalence of strictures in men vs. women and the etiology of those strictures being different, the study will focus on male subjects with single anterior urethral stricture. Subjects will be followed up post-treatment to one year and then annually for up to 5 years. The annual follow up after the first year is optional.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 18 years' old
2. Visual confirmation of stricture via cystoscopy or urethrogram
3. Single lesion anterior urethral stricture or bladder neck contracture, less than or equal to 2.0 cm
4. One to three (1-3) prior diagnosis and treatment of the same stricture (including self-catheterization) including DVIU (Direct Vision Internal Urethrotomy), but no prior urethroplasty
5. Significant symptoms of stricture such as frequency of urination, dysuria, urgency, hematuria, slow flow, feeling of incomplete emptying, recurrent UTI's.
6. IPSS score of 13 or higher
7. Lumen diameter <12F by urethrogram
8. Able to complete validated questionnaire independently
9. Qmax <10 ml/sec

Exclusion Criteria:

1. Strictures greater than 2.0 cm long.
2. Subjects that have more than 1 stricture.
3. Sensitivity to paclitaxel or on medication that may have negative interaction with paclitaxel
4. Subjects who have a suprapubic catheter and are unable to complete study required testing, such as uroflowmetry
5. Previous urethroplasty within the anterior urethra
6. Stricture due to bacterial urethritis or untreated gonorrhea
7. Stricture dilated or incised within the last 3 months
8. Presence of local adverse factors, including abnormal prostate making catheterization difficult, urethral false passage or fistula.
9. Presence of signs of obstructive voiding symptoms not directly attributable to the stricture such as BPH at the discretion of the clinical investigator
10. Previous radical prostatectomy
11. Previous pelvic radiation
12. Diagnosed kidney, bladder, urethral or ureteral stones or active stone passage in the past 6 months.
13. Diagnosed with chronic renal failure unless under hemodialysis or has a serum creatinine level greater than 2 mg/dL
14. Use of alpha blockers, beta blockers, OAB (Overactive Bladder) medication, anticonvulsants (drugs that prevent or reduce the severity and frequency of seizures), and antispasmodics where the dose is not stable. (Stable dose is defined as having the same medication and dose in the last six months.)
15. Use of Botox (onabotulinumtoxinA) in urinary system within the last 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2023-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Schorn, Study Director — Urotronic (Study Sponsor)
Locations (1):
- Libra Medical Inc, Brooklyn Park, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeLong J, Virasoro R, Pichardo M, Estrella R, Rodriguez Lay R, Espino G, Elliott S. Long-Term Outcomes of Recurrent Bulbar Urethral Stricture Treatment With the Optilume Drug-Coated Balloon: Five-Year Results From the ROBUST I Study. J Urol. 2025 Jan;213(1):90-98. doi: 10.1097/JU.0000000000004229. Epub 2024 Aug 30. PMID 39213367

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DCB Treatment
Started | 53
Completed | 29
Not Completed | 24

BASELINE CHARACTERISTICS:
Population: Intent to Treat
Arm/Group | DCB Treatment
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African Origin | 8
  Hispanic or Latino | 44
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Treatment Related Serious Complication
Description: * urethral formation of fistula
  * de novo severe urinary retention lasting > 14 consecutive days' post-treatment
  * unresolved de novo stress urinary incontinence (requiring >1 pad/day) at 90 days or earlier
  * urethra rupture or burst.
Time Frame: 90 days post-procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DCB Treatment
Number analyzed (Participants) | 53
percentage of participants | 0 [0.0 to 6.7]

2. Secondary Outcome: Stricture Recurrence Rate
Description: * IPSS score of greater than 11 at the 90-day follow-up, or
  * if a subject had a second DCB treatment (retreatment), or
  * if a subject exited the study early due to treatment failure (IPSS >11 without cystoscopically confirmed anatomical success at the time of exit or receiving additional stricture treatment with an alternative therapy).
Time Frame: 90 days post-procedure
Population: Subjects reporting 3 month IPSS outcomes or meeting the definition of treatment failure prior to the 3 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Treatment
Number analyzed (Participants) | 51
Participants | 8
Statistical Analysis 1: Comparison: DCB Treatment; Test type: Other — Recurrence < 0.5 as defined by an IPSS score of less than or equal to 11. The performance goal is met if the upper limit of the one-sided 95% confidence interval for recurrence is less than 50%; p < 0.001, 1-sample binomial z-test

ADVERSE EVENTS:
Time Frame: Adverse events were collected any time after the treatment has been initated through 5-year follow-up
Arm/Group | DCB Treatment
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 5/53
Other Adverse Events (participants affected / at risk) | 37/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCB Treatment (N=53)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Other: Fall (General disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (2)
Other: Prostatic Adenocarcinoma (Renal and urinary disorders) | 1 (1)
Myocardial Infarction, Angina, Ischemia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCB Treatment (N=53)
Dysuria (Renal and urinary disorders) | 5 (7)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Renal Colic (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 7 (8)
Urethral Stricture (Renal and urinary disorders) | 9 (11)
Hematuria (Renal and urinary disorders) | 3 (4)
Urine Flow Decreased (Renal and urinary disorders) | 3 (3)
Urethral Injuary (Renal and urinary disorders) | 1 (1)
Renal Caculi (Renal and urinary disorders) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 10 (12)
COVID-19 (Infections and infestations) | 2 (2)
Other: Orchitis (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 5 (6)
Flu-Like Symptoms (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Infusion Site Extravastation (General disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 2 (2)
Alanine Aminotransferase (Investigations) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headaches (Vascular disorders) | 3 (3)
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT03014726/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT03014726/SAP_001.pdf